CLINICAL TRIAL: NCT03827291
Title: Quantitative Observational Comparative Effectiveness of Quadratus Lumborum (QL) Block With Liposomal Bupivacaine (Exparel®) Versus Thoracic Epidural Analgesia in Patients Undergoing Laparoscopic Colectomy.
Brief Title: QL Block With Exparel in Colectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00091425
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Laparotomy; Colectomy
MeSH Terms: interventions — Tea

STUDY DESIGN:
Intervention Model Description: Compare efficacy of a quadratus lumborum block performed with liposomal bupivacaine for pain relief after laparoscopic colectomy compared to a historical cohort who received thoracic epidural analgesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Quadratus lumborum block (Experimental): Bilateral administration on each side of 30 ml aliquot containing 10 ml of liposomal bupivacaine (133 mg) and 20 ml of 0.25% bupivacaine (50 mg) in the fascial plane between the QL and psoas major muscles.
  Interventions: Drug: Exparel
- Thoracic epidural analgesia (Other): Historical cohort that received thoracic epidural analgesia.
  Interventions: Other: Thoracic epidural analgesia

INTERVENTIONS:
Drug: Exparel — Bilateral administration on each side of 30 ml aliquot containing 10 ml of liposomal bupivacaine (133 mg) and 20 ml of 0.25% bupivacaine (50 mg) in the fascial plane between the QL and psoas major muscles.
  Arms: Quadratus lumborum block
Other: Thoracic epidural analgesia — Historical cohort that received thoracic epidural analgesia
  Arms: Thoracic epidural analgesia

SUMMARY:
The purpose of this study is to determine if using a different type of injection of local anesthestic (pain medicine) in between the muscle layers of the abdominal wall (called a quadratus lumborum block) will improve pain control and be easier to manage after surgery than the current standard of care epidural (spinal injection) pain relief for patients undergoing laparoscopy colectomy.

DETAILED DESCRIPTION:
Participants in this study will receive exparel via an abdominal muscle nerve block procedure immediately prior to their operation. Participants will be in this study for 96 hours following surgery, which is typically 3 days. During participation, the study staff will review participant's electronic health records for pain scores and pain medication needs.

Participants that receive the quadratus lumborum block, may experience improved pain control and/or reduced side effects compared to the epidural pain relief option, but it is not known yet whether this will be the case.

The most common risk is being sore in the flank where the block was placed. Other risks of the block rarely occur (less than .5-1%), these can include infection, allergy to the local anesthetic, bleeding, damage to the nerve, seizures, abnormal heart rhythms, and cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective, laparoscopic colonic resection by one of three surgeons: Drs. Thacker, Mantyh or Migaly. These surgeons perform this procedure in the same manner
* Age 18-85 years
* American Society of Anesthesiologists (ASA) Physical Class I-III
* BMI 18-35 kg/m^2

Exclusion Criteria:

* Inability to consent
* Inability to speak English
* Pregnancy
* Emergency surgery
* Contraindications to regional blockade: coagulopathy or bleeding diathesis, local infection, allergy to local anesthetics
* Allergies/intolerances/contraindications to any of the multimodal agents (acetaminophen, gabapentin, ketorolac)
* Daily opioid equivalent use of 30 mg of morphine or greater at time of consent
* History of drug or alcohol abuse
* Rheumatoid arthritis
* Uncontrolled anxiety, schizophrenia or other psychiatric disorder that, in the opinion of the investigator, may interfere with the study assessments of compliance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Kumar, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Historical Controls were not considered enrolled in this study.
Groups:
- Quadratus Lumborum Block: Bilateral administration on each side of 30 ml aliquot containing 10 ml of liposomal bupivacaine (133 mg) and 20 ml of 0.25% bupivacaine (50 mg) in the fascial plane between the QL (quadratus lumborum) and psoas major muscles.
  Exparel: Bilateral administration on each side of 30 ml aliquot containing 10 ml of liposomal bupivacaine (133 mg) and 20 ml of 0.25% bupivacaine (50 mg) in the fascial plane between the QL and psoas major muscles.
Period: Overall Study
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Started | 35 | 30
Completed | 30 | 30
Not Completed | 5 | 0
Not completed — Intraoperative conversion of surgery from laparoscopic to open | 5 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [55 to 72] | 64 [50 to 71] | 63 [50 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 27 | 23 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Opioid Consumption Over 48 Hours
Description: Measured in morphine milligram equivalents.
Time Frame: From arrival to PACU to 48 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 30 | 30
morphine milligram equivalents | 33 [8 to 76] | 61 [40 to 85]

2. Secondary Outcome: Pain While Coughing as Measured by 11-point Numeric Rating Scale (NRS-11)
Description: The NRS-11 is an 11-point scale where 10=worst pain imaginable and 0= no pain.
Time Frame: 30 minutes after arrival to Post-Anesthesia Care Unit (PACU), and at 8 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours and 168 hours post Exparel administration
Population: Data not collected at 144 hours or 168 hours.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 30 | 30
score on a scale
  30 minutes | 5 [3 to 7] | 4 [0 to 7]
  8 hours | 3 [2 to 6] | 0 [0 to 3]
  24 hours | 3 [2 to 4] | 2 [0 to 4]
  36 hours | 2 [0 to 4] | 2 [0 to 4]
  48 hours | 4 [2 to 5] | 3 [0 to 7]
  72 hours | 2 [1 to 5] | 3 [0 to 6]
  96 hours | 2 [0 to 5] | 5 [3 to 6]
  120 hours | 2 [1 to 5] | 5 [2 to 5]
  144 hours: number analyzed (Participants) | 0 | 0
  168 hours: number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Number of Participants With Block Success
Description: Presence of demonstrable sensory block over 4 points on the abdomen (one in each of the 4 quadrants), as tested by response to pinprick. Subjects will be asked to report whether the stimulus feels "sharp" or "dull", indicating block failure and success respectively.
Time Frame: 30 minutes after arrival to PACU, 8 hours, 24 hours, 36 hours, 48 hours and 72 hours post Exparel administration
Measure: Count of Participants; unit: Participants
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 30 | 30
Participants | 7 | 1

4. Other Pre Specified Outcome: Number of Participants With Adverse Events Related to the Block
Description: Subjects will be evaluated for potential adverse events related to the block including evidence of hematoma, infection, unexpected sensory or motor deficit, local anesthetic systemic toxicity, as well as transient weakness of the hip flexor muscles (a known possible side-effect of QL block).
Time Frame: From administration of Exparel through 168 hours post Exparel administration
Measure: Count of Participants; unit: Participants
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 30 | 30
Participants | 6 | 8

5. Other Pre Specified Outcome: Satisfaction With Postoperative Pain Control
Description: Overall subject satisfaction with pain control will be recorded on an 11-point scale: 10=highly satisfied, 0=completely unsatisfied.
Time Frame: Up to 48 hours post Exparel administration
Population: Not applicable to the historical thoracic epidural analgesia group.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 30 | 0
score on a scale | 8 [3 to 9] |

6. Other Pre Specified Outcome: Hospital Length of Stay
Description: Measured both by raw length of stay and by time to achieving "discharge readiness", defined by the presence of 3 criteria: a pain score of 3 or less with ambulation, no opioids required in the preceding 6 hours, and the ability to perform self-care (go to the toilet, dress, and shower).
Time Frame: From administration of Exparel through hospital discharge
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 30 | 30
hours | 27 [24 to 46] | 55 [52 to 97]

7. Other Pre Specified Outcome: Number of Participants With Opioid-related Adverse Events
Description: Adverse events include nausea, vomiting, ileus, constipation, orthostasis, pruritis, urinary retention, respiratory depression.
Time Frame: From administration of Exparel through 168 hours post Exparel administration
Measure: Count of Participants; unit: Participants
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 30 | 30
Participants | 10 | 19

8. Other Pre Specified Outcome: Time to First Mobilization
Time Frame: From time of arrival in PACU through first mobilization
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 30 | 30
hours | 15 [8 to 19] | 31 [27 to 49]

9. Other Pre Specified Outcome: Cost
Description: Hospital costs including pharmacy-related costs, costs due to opioid-related adverse events, the cost associated with nursing interventions and drugs to treat opioid-related adverse events, and overall hospital admission costs will be calculated.
Time Frame: From time of arrival in PACU through 96 hours post Exparel administration
Population: Data not collected.
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Sleep Quality as Measured by Two Questions
Description: Each question has a scale of 0 (no interference) to 10 (completely interferes) and the two scores are averaged: "How much did pain interfere with falling asleep?", "How much did pain interfere with staying asleep?"
Time Frame: Up to 168 hours post Exparel administration
Population: Not applicable to the historical thoracic epidural analgesia group.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
Number analyzed (Participants) | 30 | 0
score on a scale | 4 [2 to 8] |

ADVERSE EVENTS:
Time Frame: From arrival to PACU to postoperative day 7
Arm/Group | Quadratus Lumborum Block | Thoracic Epidural Analgesia
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 10/30 | 19/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quadratus Lumborum Block (N=30) | Thoracic Epidural Analgesia (N=30)
Extended hospital stay due to left lower extremity numbness (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quadratus Lumborum Block (N=30) | Thoracic Epidural Analgesia (N=30)
Hypotension (Cardiac disorders) | 0 | 8
Orthostasis (Cardiac disorders) | 3 | 8
Pruritis (Nervous system disorders) | 1 | 6
Urinary retention (Renal and urinary disorders) | 1 | 4
Unexpected sensory deficit (Nervous system disorders) | 6 | 3
Hip flexor weakness (Nervous system disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 10 | 19
Vomiting (Gastrointestinal disorders) | 3 | 8
Constipation (Gastrointestinal disorders) | 3 | 2
Ileus (Gastrointestinal disorders) | 1 | 4
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03827291/Prot_SAP_000.pdf